CLINICAL TRIAL: NCT01050868
Title: Comparison of the Management of Post-prandial Hyperglycemia by Multiple Bolus Calculators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RD000811
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (1):
- Single Arm (Experimental)
  Interventions: Device: Accu-Chek Combo Kit mg DE/de

INTERVENTIONS:
Device: Accu-Chek Combo Kit mg DE/de

SUMMARY:
This prospective, non-randomized, non-controlled, interventional study will determine whether the Roche automated bolus caclulator (ABC) reduces post-meal hyperglycemia better than the competitor's ABC without causing significant hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects >/= 18 years at screening
* Type 1 diabetics currently using an insulin pump for management of their diabetes and have been on a pump for at least at least 6 months prior to the screening visit
* Subjects have to use a fast acting analog insulin
* HbA1c = 9% (measured with DCA 2000)
* Willing to perform periods of intensive blood glucose (BG) monitoring for up to 21 days prior to the study (~10 tests per day) with skipped meals and testmeals
* Willing to use the 3 different bolus calculators during the course of the study
* Willing to undergo planned hyperglycemia
* Willing to perform high frequency BG monitoring (> 20 / day) during the experiment

Exclusion Criteria:

* Type 2 Diabetes
* Manifest severe late complications of diabetes (e.g. severe macro- or microangiopathy, severe neuropathy, severe retinopathy and/or severe nephropathy)
* Current addiction to alcohol or substances of abuse
* Pregnant or lactating women
* Any known life-threatening disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To compare the difference between the self-monitoring blood glucose (SMBG) value achieved at 6 hours after meals with induced post-prandial hyperglycemia and the mean target value of 110 mg/dL. Target post-prandial range is 80-140 mg/dL. | 6 hours after meal

SECONDARY OUTCOMES:
To compare the absolute difference between the SMBG value and the target value between the calculators | 6 hours after meal
To compare theto compare the relative difference (multiplied by 100) between the SMBG value and the target value between the calculators | 6 hours after meal
To compare the absolute relative difference (RAD, multiplied by 100) between the SMBG value and the target value between the calculators | 6 hours after meal

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Petersen, Study Director — Roche Diagnostics GmbH / Diabetes Care
Locations (1):
- Ulm, Germany